# **EAACI Interest Group on Insect Venom Hypersensitivity**

# STUDY PROTOCOL

# **EADOAS-Study**

The <u>effect</u> of <u>antihypertensive</u> <u>drugs on severity of <u>anaphylaxis</u> and <u>side</u> –effects during venom immunotherapy EAACI multicenter study</u>

## NCT04269629

# **Study coordinator:**

Gunter J. Sturm, MD, PhD
Department of Dermatology
Medical University of Graz
Auenbruggerplatz 8
8036 Graz, Austria

Telephone: +43-650-5142129 Telefax: +43-316-385-12466

E-mail: gunter.sturm@medunigraz.at

# **Table of Contents**

| 1. | S | tud | y syn | opsis | 4 |
|---|---|---|---|---|---|
| 2. | Ir | ndic | atior | n and objectives | 6 |
| | 3.1 | | Beta | -blockers | 6 |
| | 3 | .1.1 | | Background | 6 |
| | 3 | .1.2 | | Potential effect on immunotherapy | 7 |
| | 3 | .1.3 | | Current recommendations | 8 |
| | 3.2 | | ACE- | -inhibitors | 8 |
| | 3 | .2.1 | · | Background | 8 |
| | 3 | .2.2 | | Potential effect on immunotherapy | 8 |
| | 3 | .2.3 | | Current recommendations | 9 |
| 4. | Ju | ustif | ficati | on of the study | 9 |
| 5. | S | tud | y crit | eria | LO |
| | 5.1 | | Prim | ary objective | LO |
| | 5.2 | | Seco | ondary objectives | LO |
| 6. | Р | atie | nts a | and methods | LO |
| | 6.1 | | Subj | ect eligibility | LO |
| | 6.2 | | Inclu | usion criteria | LO |
| | 6.3 | | Excl | usion criteria for phase 2 (no exclusion criteria for phase 1) 1 | LO |
| | 6.4 | | Met | hods | ۱1 |
| | 6 | .4.1 | | Personal history | l1 |
| | 6 | .4.2 | | Laboratory tests | l1 |
| | 6 | .4.3 | , | Skin testing (Intradermal skin test and/or prick testing) | l1 |
| | 6 | .4.4 | | Venom immunotherapy (VIT) | l1 |
| 7. | О | ver | all st | udy design and plan | L2 |
| 8. | S | che | dule | of study procedures | L2 |
| 9. | Ε | arly | tern | nination of study1 | L3 |
| 10 | | Da | ıta re | ecording and documentation | L3 |
| 11 | | Sta | atisti | cal methods | L3 |
| 12 | | Re | gula | tory and ethical obligations1 | L5 |
| | <b>12.</b> 1 | L | Insti | tutional Review Board 1 | L5 |
| | 12.2 | 2 | Info | rmed consent | L5 |
| | 12.3 | 3 | Stud | ly initiation1 | L5 |
| | 12.4 | 1 | Case | report forms | 15 |

| 13. | Table | S | |
|-----|--------|-----------|----|
| 13 | .1 Tak | ole 1 | 16 |
| | | Table 1A | |
| | 13.1.2 | Table 1B | 16 |
| 13 | .2 Tak | ole 2 | |
| | | eviations | |
| | | ences | |

# 1. Study synopsis

| ADDITCANT / Cuntor Sturm MD DbD | |
|---|---|
| Gunter J. Sturm, MD, PhD | |
| COORDINATING Department of Dermatology | |
| INVESTIGATOR Medical University of Graz | |
| Auenbruggerplatz 8 | |
| 8036 Graz, Austria | |
| Telephone: +43-650-5142129 | |
| Telefax: +43-316-385-12466 | |
| E-mail: <a href="mailto:gunter.sturm@medunigraz.at">gunter.sturm@medunigraz.at</a> | |
| TITLE OF STUDY The effect of antihypertensive drugs on severity of anaphylax | is and |
| side-effects during venom immunotherapy | |
| SHORT TITLE EADOAS-Study | |
| POPULATION Patients with a history of anaphylactic sting reaction | |
| OBJECTIVE(S) The primary objective of this study is to evaluate whether | subjects |
| under antihypertensive treatment with beta-blockers and | or ACE- |
| inhibitors show more side effects during VIT compared to | subjects |
| with no antihypertensive treatment. | |
| INTERVENTION(S) Venom immunotherapy (VIT) | |
| KEY INCLUSION AND <u>Inclusion criteria:</u> Subjects aged from 35 to 85 years with a h | istory of |
| <b>EXCLUSION CRITERIA</b> anaphylactic sting reaction | |
| Exclusion criteria (only for phase 2): Absolute contraindica | tions for |
| VIT, Pretreatment with Omalizumab | |
| OUTCOME(S) Proportion of side-effects during venom immunotherapy | |
| STUDY TYPE Prospective multicenter observational study | |
| STATISTICAL ANALYSIS The primary analysis will compare the proportion of objective | side |
| effects between the groups (subjects under antihypertensive | |
| treatment vs. subjects without antihypertensive treatment) ( | ising a |
| Mantel-Haensel estimate of the odds ratio stratified by clinic | Ŭ |
| A logistic regression model will be used to central for other n | accibla |
| A logistic regression model will be used to control for other p | ossible |
| confounders | |
| ETHICAL APPROVALS Participating study centers have to obtain ethical approvals for | rom |
| their institutional review boards. | |
| SPONSORING Unrestricted grants from pharmaceutical companies | |
| SAMPLE SIZE 1319 | |
| TRIAL DURATION July 1, 2014 – December 31, 2019 | |
| (End of inclusion phase: January 31, 2018) | |

| PARTICIPATING | Name | Address | Country |
|---|---|---|---|
| CENTERS | Prof. Gunter J Sturm,<br>MD, PhD | Department of Dermatology Medical University of Graz | Austria |
| | | Auenbruggerplatz 8<br>8036 Graz, Austria | |
| | Prof. Norbert Reider, | Clinical Department of | Austria |
| | MD | Dermatology | . 10.001.10 |
| | | Medical University of | |
| | | Innsbruck | |
| | | Anichstraße 35 | |
| | | 6020 Innsbruck, Austria | |
| | Thomas Hawranek, MD | Department of Dermatology | Austria |
| | | SALK<br>Paracelsus Medical | |
| | | University Salzburg | |
| | | Müllner Hauptstraße 48 | |
| | | 5020 Salzburg, Austria | |
| | Prim. UnivDoz. Georg | Department of Dermatology | Austria |
| | Klein, MD | Elisabethinen Hospital Linz | |
| | | Fadingerstrasse 1 | |
| | D. D. Cl. C. Willed | 4020 Linz, Austria | A -1 - |
| | PrivDoz. Stefan Wöhrl, | Floridsdorf Allergy Center<br>Franz-Jonas-Platz 8/6 | Austria |
| | IVID | 1210 Vienna, Austria | |
| | Prof. Christof Ebner, MD | Ambulatory for Allergy and | Austria |
| | , | Clinical Immunology - AAKI | |
| | | GmbH | |
| | | Reumannplatz 17 | |
| | | 1100 Vienna, Austria | |
| | List to be continued | | |
| SPONSORING | Unrestricted grants from pharmaceutical companies | | |

#### 2. Indication

There is an ongoing debate whether antihypertensive treatment with beta-blockers and/or ACE-inhibitors comprises a risk factor for more severe anaphylactic reactions due to insect stings. Side effects under venom immunotherapy (VIT) could be more severe and more frequent. In the literature, data are controversial and originate from case reports or statistically underpowered studies.

#### 3. Introduction

Since the introdution of beta-blockers in the early 1960s and the availability of ACE-inhibitors in the early 1980s, there is an ongoing discussion about negative effects of those substances on allergic reactions and side-effects during allergen immunotherapy. Although there is a theoretical and anectotal clinical evidence for possible interactions, data of studies are controversial and their role as risk factors is a debated issue. All available studies have drawbacks and are underpowered. Therefore, current recommendations are practice-oriented but not sufficiently evidence-based. To stop the endless debate, a well planned multicenter study ist needed.

#### 3.1 Beta-blockers

Beta-blockers are mostly used to treat arterial hypertension and are valuable drugs in the treatment of cardiovascular disease. However, they are also prescribed for non-cardiac conditions like migraine prophylaxis or symptomatic treatment of skeletal muscle tremor.

## 3.1.1 Background

Four main types of adrenergic receptors ( $\alpha_1$ ,  $\alpha_2$ ,  $\beta_1$ ,  $\beta_2$ ) can be roughly distinguished according to their affinity to norepinephrine and epinephrine. In brief, stimulation of  $\beta_1$  receptors induces a positive chronotropic and inotropic effect on the heart as well as a renin release of the kidney.  $\beta_2$  stimulation results in dilatation of blood vessels and bronchioles, and  $\alpha_2$  stimulation induces contraction of blood vessels and bronchioles  $^1$ . Basically,  $\beta$  blockade inhibits the effect of both endogenously released and therapeutically administered epinephrine on  $\beta$  receptors in case of anaphylaxis. Therefore epinephrine treatment can be ineffective or due to the block of  $\beta_1$  and  $\beta_2$  actions may facilitate unopposed  $\alpha$ -adrenergic effects like bronchoconstriction and bradycardia  $^2$ .

#### 3.1.2 Potential effect on immunotherapy

- Side effects do not appear to be more frequent, but maybe more serious

- Side effects could be refractory to treatment
- Emergency treatment may cause paradoxical treatment effects

Both beta blockers and allergen immunotherapy are frequently prescribed, therefore allergists commonly encounter patients who are candidates for immunotherapy and are treated with beta blockers. Fatality studies have shown that particularly elderly patients with pre-existing cardiovascular disease die from hymenoptera venom allergy<sup>3</sup>. Therefore unlike for respiratory allergies, immunotherapy with hymenoptera venoms is commonly performed in elderly patients who are more likely to be on beta blocker treatment.

The risk of beta blocker treatment is still questionable. There is plenty of experimental human<sup>4, 5</sup> and animal studies<sup>6-8</sup> mainly performed in the 1970s and 80s as well as anecdotal clinical evidence<sup>9-15</sup> that anaphylaxis may be influenced by pharmacodynamics of βblockade. In theory,  $\beta$ -blockade perturbs the control of endogenously produced mediators of anaphylaxis resulting in an enhanced generation, release, and reduced effects of these mediators on the end organs<sup>2</sup>. If anaphylaxis occurs in a patient on beta-blocker, it may therefore be more severe and protracted. There is also evidence that even beta-blocker eye drops have systemic effects<sup>16-19</sup>. However, the plurality of uncontrolled variables makes the susceptibility of individual patients to this effect of topically and orally applied beta-blockers largely unpredictable<sup>2</sup>. The second point is that emergency treatment with epinephrine may be ineffective or promote undesired  $\alpha$ -adrenergic and vagotonic effects<sup>20</sup>.  $\beta$ -blockade dramatically alters pharmacotherapeutic actions of epinephrine and isoproterenol, as up to 80-fold higher doses may be necessary<sup>5, 21</sup>. Additionally, the block of  $\beta_1$  and  $\beta_2$  actions of epinephrine may facilitate unopposed  $\alpha$ -adrenergic and reflex vagonotic effects, which can result in increased mediator release, bronchoconstriction and bradycardia<sup>5</sup>. The pronounced α-receptor activation in the presence of epinephrine may also constrict coronary arteries or exaggerate systemic pressor effects of epinephrine leading to severe hypertensive episodes.

There are three clinical studies dealing with the question whether patients taking beta-blockers are at increased risk of having side effects during immunotherapy. Hepner et al<sup>22</sup> prospectively studied 3178 patients; 68 patients were taking beta-blockers. Although statistically 3 patients were expected to have systemic reactions, only one patient taking a beta-blocker had a systemic reaction. In a retrospective study of Mueller et al<sup>23</sup>, 1389 patients were included, and 25 patients were on beta-blockers during immunotherapy. They also did not find an increased incidence of systemic reactions, and reactions were not more severe than in the control group. Most recently, an EAACI observational prospective multicenter study on 680 patients (15 on beta-blockers) could not identify beta-blocker therapy as independent predictor for an emergency intervention<sup>24</sup> during immunotherapy. Interestingly, in a former EAACI observational study on 962 patients<sup>25</sup> (52 on beta-blockers) beta blocker were not identified as independent risk factor for severe anaphylaxis, which

was consistent with a large Australian study<sup>26</sup>. In this study, case records of 1149 patients were retrospectively analyzed. Univariate analyses suggested that reaction severity was influenced by beta-blockers. However, in the multivariate analysis beta-blockers were not identified as independent risk factor. Recently, 657 patients suitable for VIT were included in a large single-center observational study. 59 were on beta-blocker treatment; 27 on both, ACE-inhibitors and beta blockers. Again, beta blockers were not identified to be correlated with severe anaphylaxis<sup>27</sup>. More recently, again controversial data have been published: Beta-blockers were not associated with severe anaphylactic symptoms such as syncope or hypotension, but with 3 or more organ involvement and hospitalization<sup>28</sup>.

#### 3.1.3 Current recommendations

There is good evidence in the literature that anaphylaxis is not more frequent in patients receiving beta-blockers. On the other side patients may be at increased risk from more severe systemic reactions and from ineffective emergency treatment. Therefore there is still a relative contraindication for beta blockers in subjects allergic to hymenoptera venom.

#### 3.2 ACE-inhibitors

ACE-inhibitors are primarily used to treat arterial hypertension and congestive heart failure.

#### 3.2.1 Background

The renin angiotensin aldosterone system (RAS) regulates blood pressure. The system in general increases blood pressure by reduced salt and water excretion and vasoconstriction if blood pressure acutely drops<sup>1</sup>. ACE inhibitors block conversion of angiotensin I to angiotensin II, which results in vasodilatation and reduced blood volume. Therefore, hypotension during anaphylaxis may not sufficiently counteracted by the inhibited RAS.

#### 3.2.2 Potential effect on immunotherapy

- Diminished ability to counteract allergy-induced hypotension

There is some anecdotal clinical evidence that a subset of patients receiving venom immunotherapy tend to have more serious hypotension in case of side effects<sup>29, 30</sup>. In theory, the RAS is part of the compensatory physiologic response to anaphylaxis and thus ACE-inhibitors may hamper an effective response in some instances of anaphylaxis. However, also a dysfunctional RAS in which overall RAS activity is diminished might aggravate symptoms due to an insufficient response to anaphylaxis<sup>31-33</sup>.

The role of ACE-inhibitors as risk factor for more severe anaphylaxis is still a debated issue. In a large Australian retrospective analysis done by Brown<sup>26</sup>, 1149 patients who have had anaphylaxis were included. Among these, fifty-seven patients were on ACE-inhibitor treatment. Multivariate analysis did not identify ACE-inhibitors as independent risk factor. However, in an EAACI observational prospective multicenter study on 962 patients with hymenoptera allergy, the 42 patients receiving ACE inhibitors had an approximately 2.3-fold increased risk for severe anaphylaxis (odds ratio 2.26, 95% CI 1.13 - 4.56) <sup>25</sup>.

The second EAACI observational multicenter study on 680 VIT patients (18 patients on ACE-inhibitors) did not identify ACE-inhibitors as independent risk factor for side effects.

Recently, 657 patients suitable for VIT were included in a large single-center observational study. 32 were on ACE and 27 on beta-blocker treatment. Again, ACE-inhibitors were not identified to be correlated with severe anaphylaxis<sup>27</sup>. Another retrospective analysis revealed that ACE-inhibitors were not associated with severe anaphylactic symptoms such as syncope or hypotension, but with 3 or more organ involvement and hospitalization<sup>28</sup>. Most recently, in a study on 743 patients (thereof 90 on ACE inhibitor treatment) ACE inhibitors did not increase the frequency of side-effects during the buildup phase of VIT<sup>34</sup>.

#### 3.2.3 Current recommendations

If ACE-inhibitors increase the risk of more serious anaphylaxis is still a debated issue. Currently, the recommendation that patients receiving ACE-inhibitors are more likely to have side effects during immunotherapy is only based on case reports. Nevertheless, until there will not be new evidence, current guidelines recommend to replace ACE-inhibitors, if feasible.

# 4. Justification of the study

Although a considerable number of studies on this topic were performed, all studies were underpowered to identify beta blockers and/or ACE inhibitors as risk factors. The number of included patients was usually high; however, the proportion of patients on antihypertensive treatment was low ranging from 2-11%<sup>22, 34</sup>. In the current study we plan to enroll 1319 patients aged 35-85. Considering retrospective data from our own institution it is assumed that 24% (317) will be on beta blockers and/or ACE inhibitors. Based on these data, a clear statement on the risk of antihypertensive treatment will be possible.

#### 5. Study criteria

## 5.1 Primary objective

• The primary objective of this study is to evaluate whether subjects under antihypertensive treatment with beta-blockers and/or ACE-inhibitors show more side effects during VIT compared to subjects with no antihypertensive treatment.

# 5.2 Secondary objectives

- To evaluate whether subjects under antihypertensive treatment with beta-blockers and/or ACE-inhibitors have more severe sting reactions.
- To correlate the prevalence of cardiovascular diseases and/or hypertension with the risk for more severe systemic sting reactions and with more severe and more frequent side effects under VIT.
- To evaluate whether bee venom is associated with a higher frequency of side-effects.
- To evaluate whether high sigE levels are correlated to a higher frequency of side-effects.
- To evaluate whether high tryptase levels are correlated to a higher frequency of sideeffects.
- To evaluate whether quicker up-dosing protocols are correlated to a higher frequency of side-effects.
- To evaluate efficacy of VIT by sting challenges or field stings and look for differences between patients with and without antihypertensive treatment

#### 6. Patients and methods

#### 6.1 Subject eligibility

Patient selection takes place on the basis of the inclusion and exclusion criteria

#### 6.2 Inclusion criteria

- Legally competent male and female individuals aged from 35 to 85 years with a history of systemic sting reaction (≥ grade I according to the classification by Ring and Messmer, Table 1).
- Age ≥35 and ≤85 years

# 6.3 Exclusion criteria for phase 2 (no exclusion criteria for phase 1)

- Absolute contraindications for VIT
- Pretreatment with Omalizumab

#### 6.4 Methods

## 6.4.1 Personal history

6.4.2 Personal history is recorded at Visit 1 if patients have met inclusion and exclusion criteria. Previous sting reactions, allergies, diseases and current medication will be recorded in the CRF.

Symptoms will be divided into subjective and objective symptoms. <u>Subjective symptoms are</u>: feeling of warmth, isolated pruritus, headache, general fatigue, anxiety, dysphagia, throat tightness, chest tightness, nausea, vertigo, perception of impending doom

<u>Objective symptoms are</u>: flush, urticarial, angioedema, dyspnea, hoarseness, drop in blood pressure, tachycardia, vomiting, abdominal cramping, bronchospasm, involuntary urination, involuntary defecation, loss of consciousness, cardiac arrest, apnoea

#### 6.4.3 Laboratory tests

Total and specific IgE (bee and vespid venom, rApi m 1, rVes v 1, rVes v 5) as well as serum tryptase will be determined.

Measurements will be performed as part of clinical routine procedures by ImmunoCAP® (Thermo Fisher Scientific, Waltham, MA, USA), according to the manufacturer's instructions.

## 6.4.4 Skin testing (Intradermal skin test and/or prick testing)

Skin testing is performed routinely within the standard diagnostic procedure of each center.

# 6.4.5 Venom immunotherapy (VIT)

There is no standard buildup phase; centers use their own standard protocols. Typically, conventional (outpatient), Cluster/Ultrarush- (partial inpatient) and Rush-protocols (inpatient) will be performed. The respective venom that is used for VIT will be recorded (bee or wasp venom, trade name, company). Injections will be administered subcutaneously in the dorsal part of the upper arm, one hand's breadth above the elbow, or in the volar part of the thigh. All interventions will be performed according to the in-house protocols of participating centers.

#### 7. Overall study design and plan

The study is conducted as an open, prospective observational study on an outpatient basis. After giving the Informed Consent subjects will be screened at Visit 1. Subjects meeting the inclusion and exclusion criteria will be included (phase 1). If subjects agree to receive VIT, side effects during the buildup phase will be recorded (phase 2). At the first annual control visit side effects during maintenance phase and, if applicable, the outcome of field stings of sting challenge tests will be recorded (phase 3). No additional study-related visits are required.

Participation in this study will have no influence on decision-making for venomimmunotherapy. All procedures have to be in concordance with current EAACI guidelines<sup>35, 36</sup> and will be conducted individually by each study center.

Detailed schedule of events please see Table 2.

# 8. Schedule of study procedures

#### Phase 1 (Screening, inclusion) – Visit 1. (week 0)

The following procedures will be performed:

- Ask the subject to read and sign the Informed Consent
- Review of inclusion and exclusion criteria
- Collect medical and allergy history, recording of co-medication
- Collect demographics
- Perform skin testing and determination of IgE and serum tryptase (CAP)
- Record decision regarding venom immunotherapy (yes/no)

# Phase 2 (up-dosing of VIT) – Visit 2. (0-4 weeks after reaching maintenance dose)

- Re-collect medical history, recording of co-medication
- Record of up-dosing scheme and of the respective venom used for VIT
- Record pre-treatment during VIT
- Record of side-effects during VIT up-dosing

# Phase 3 (maintenance phase) – Visit 3/3a (at least 12 months [+/- 2 months] after reaching maintenance dose)

- Re-collect medical history, recording of co-medication
- Record of side-effects during VIT maintenance phase

## Phase 3 (maintenance phase) – Visit 3b/3c optional

- Document field stings and sting challenges
- Record outcome of field sting or sting challenge

## 9. Early termination of study

The subject will be advised in the Informed Consent Form that he/she has the right to withdraw from the trial at any time without prejudice. Reasons for a premature treatment stop will be documented, if feasible.

The enrolment of new subjects will be suspended if more than 5 serious anaphylactic reactions (≥grade III according to Ring & Messmer; except bronchoconstriction) during buildup phase in patients with antihypertensive treatment occur.

#### 10. Data recording and documentation

Data are recorded in case report forms (CRFs). Data will also be collected using a web based form. Data regarding this study is recorded, analyzed, and archived in anonymized form.

#### 11. Statistical methods

All patients who participate in this study belong to one of the following two groups for the analyses: the group without antihypertensive medication, and the group on antihypertensive medication (beta blockers and/or ACE inhibitors). The analyses will be based on the patients who completed buildup phase of immunotherapy.

Categorical variables will be described with percentages, and continuous variables will be expressed as means ± standard deviation or median with interquartile range.

Statistical analysis will be performed using IBM SPSS Statistics 21. A 5% level of significance will be used throughout. In all analyses, an appropriate transformation may be used to obtain approximate normality.

## 11.1 Analysis of primary endpoint

The primary endpoint for the study is the presence of objective side effects during immunotherapy which is defined as binary outcome: yes if any grade of objective side effect occurred, no otherwise.

The primary analysis will compare the proportion of objective side effects between the groups using a Mantel-Haensel estimate of the odds ratio stratified by center. A logistic regression model will be used to control for other possible confounders: age, gender, cardiovascular disease, hypertension, chronic bronchial disease or asthma, total IgE, venom-specific IgE, tryptase levels, mastocytosis, skin test reactivity, and study centers.

# 11.2 Analysis of secondary endpoints

For the analysis of secondary endpoints, comparison between groups will be made by using  $\chi 2$  statistics or the Fisher exact test for categorical variables and by t-test or the Mann-Whitney U test for continuous variables.

# 11.3 Sample size

It is assumed that 24% of the patients will be on beta blockers and/or ACE inhibitors. A  $\chi 2$  test with a two-sided 5% significance level has a 80% power to detect the difference between the group without antihypertensive medication with 6% side effects during VIT and the group on beta blockers and/or ACE inhibitors with 12.3% side effects during VIT (OR = 2.2) when the sample sizes are 631 and 200 (a total sample size of 831), respectively.

The drop-out rate includes study dropouts (30%) who do not start immunotherapy and study dropouts (10%) who do not end immunotherapy. This results in a drop-out rate of 37% and a required number of 1319 patients.

## 12. Regulatory and ethical obligations

#### 12.1 Institutional Review Board

Each study center will follow the respective regulations of the local ethical review board. Approval of the study seems necessary particularly with respect to the statistical evaluation of patient data, which have to be processed in an anonymized form. Only routine diagnostic procedures will be performed. No additional diagnostic test, treatment or check of efficacy with sting challenges will be done solely for the study

# 12.2 Informed consent

Informed consent has to be obtained from each patient before inclusion in the study. The local policies have to be followed. Translations to the national language have to be done by study centers. Informed consent has to be documented. The documentation will remain with the study documents throughout the study, and must be available for inspection by any authorized personnel.

## 12.3 Study initiation

The following documents must be on file at the study sites before the start of this study:

- Current curricula vitae of all investigators involved in the study
- Documentation of Institutional Review Board approval of the following:
  - Protocol with version number and date, and date of approval
  - Informed Consent Form with version number and date, and date of approval

## 12.4 Case report forms

The study coordinator will supply copies of the forms. A center code will be assigned to each study center. Consecutive patients receive consecutive numbers by the study center. The anonymization key is kept together with the patients' written informed consent at each center. Data of each paper-CRF will be entered into an online e-CRF form in anonymised form. The originals are kept in the center.

# 13. Tables

# 13.1 Table 1

# 13.1.1 Table 1A

Classification of systemic reactions modified according to J. Ring and Messmer  $^{35,\,37}$ 

| Cradal | Generalised skin symptoms (e.g. flush, generalised urticaria, |
|---|---|
| Grade I | angioedema) |
| Grade II | Mild to moderate pulmonary, cardiovascular (tachycardia, hypotension, |
| Grade II | dizziness), and/or gastrointestinal symptoms (nausea) |
| Grade III | Anaphylactic shock, loss of consciousness, life-threatening spasm of |
| Grade III | smooth muscles (bronchi, uterus, etc.) |
| Grade IV | Cardiac and/or respiratory arrest |

# 13.1.2 Table 1B

Classification of systemic reactions according to Mueller<sup>38</sup>

| Grade I | Generalised urticaria, itching, malaise and anxiety |
|---|---|
| | Any of the above plus two or more of following: |
| Grade II | Generalised oedema; constriction in chest; wheezing; abdominal pain, |
| | nausea and vomiting; and dizziness. |
| | Any of the above plus two or more of following: |
| Grade III | Dyspnea; dysphagia; hoarseness or thickened speech; confusion; and |
| | feeling of impending disaster. |
| | Any of above plus two or more of following: |
| Grade IV | Cyanosis; fall in blood pressure; collapse incontinence; and |
| | unconsciousness. |

# 13.2 Table 2

| Study procedures | Visit 1 Screening/Inclusion | Visit 2<br>Up-dosing | Visit 3/3a Maintenance Phase | Visit 3b/c <sup>a</sup> Field sting / sting challenge |
|---|---|---|---|---|
| Informed consent | X | | | |
| Inclusion/Exclusion review | Х | | | |
| Allergy history | x | | | |
| Medical history / co-<br>medication | Х | X | Х | х |
| Demographics | x | | | |
| Collect results of IDT and CAP | Х | | | |
| Recording of decision regarding venom immunotherapy (yes/no) | Х | | | |
| Recording of venom used for VIT | | Х | | |
| Recording of side-effects | | Х | Х | |
| Recording of stinging insect | | | | х |
| Recording of sting reaction | | | | Х |

<sup>&</sup>lt;sup>a</sup> if applicable.

# 14. Abbreviations

ACE angiotensin converting enzyme

CAP ImmunoCAP® (test for sIgE determination)

CI confidence interval

CRF case report form

EAACI European Academy of Allergology and Clinical Immunology

IDT intradermal test

OR odds ratio

RAS renin angiotensin (aldosterone) system

sIgE specific IgE antibodies

tlgE total lgE

VIT venom immunotherapy

#### 15. References

1. Silbernagel S, Despopoulos A. Color Atlas of Physiology. 6th ed. New York (NY): Thieme Publishing Group; 2009.

- 2. Toogood JH. Beta-blocker therapy and the risk of anaphylaxis. CMAJ 1987; 137:587-8, 90-1.
- 3. Sasvary T, Muller U. [Fatalities from insect stings in Switzerland 1978 to 1987]. Schweiz Med Wochenschr 1994; 124:1887-94.
- 4. Shereff RH, Harwell W, Lieberman P, Rosenberg EW, Robinson H. Effect of beta adrenergic stimulation and blockade on immediate hypersensitivity skin test reactions. J Allergy Clin Immunol 1973; 52:328-33.
- 5. Hiatt WR, Wolfel EE, Stoll S, Nies AS, Zerbe GO, Brammell HL, et al. beta-2 Adrenergic blockade evaluated with epinephrine after placebo, atenolol, and nadolol. Clin Pharmacol Ther 1985; 37:2-6.
- 6. Assem ES, Schild HO. Antagonism by beta-adrenoceptor blocking agents of the antianaphylactic effect of isoprenaline. Br J Pharmacol 1971; 42:620-30.
- 7. Matsumura Y, Tan EM, Vaughan JH. Hypersensitivity to histamine and systemic anaphylaxis in mice with pharmacologic beta adrenergic blockade: protection by nucleotides. J Allergy Clin Immunol 1976; 58:387-94.
- 8. Nisam MR, Zbinden A, Chesrown S, Barnett D, Gold WM. Distribution oand pharmacological release of histamine in canine lung in vivo. J Appl Physiol 1978; 44:455-63.
- 9. Madowitz JS, Schweiger MJ. Severe anaphylactoid reaction to radiographic contrast media. Recurrences despites premedication with diphenhydramine and prednisone. JAMA 1979; 241:2813-5.
- 10. Jacobs RL, Rake GW, Jr., Fournier DC, Chilton RJ, Culver WG, Beckmann CH. Potentiated anaphylaxis in patients with drug-induced beta-adrenergic blockade. J Allergy Clin Immunol 1981; 68:125-7.
- 11. Newman BR, Schultz LK. Epinephrine-resistant anaphylaxis in a patient taking propranolol hydrochloride. Ann Allergy 1981; 47:35-7.
- 12. Berkelman RL, Finton RJ, Elsea WR. Beta-adrenergic antagonists and fatal anaphylactic reactions to oral penicillin. Ann Intern Med 1986; 104:134.
- 13. Hamilton G. Severe adverse reactions to urography in patients taking beta-adrenergic blocking agents. Can Med Assoc J 1985; 133:122.
- 14. Javeed N, Javeed H, Javeed S, Moussa G, Wong P, Rezai F. Refractory anaphylactoid shock potentiated by beta-blockers. Cathet Cardiovasc Diagn 1996; 39:383-4.
- 15. Kivity S, Yarchovsky J. Relapsing anaphylaxis to bee sting in a patient treated with beta-blocker and Ca blocker. J Allergy Clin Immunol 1990; 85:669-70.
- 16. Diggory P, Heyworth P, Chau G, McKenzie S, Sharma A, Luke I. Improved lung function tests on changing from topical timolol: non-selective beta-blockade impairs lung function tests in elderly patients. Eye (Lond) 1993; 7 ( Pt 5):661-3.
- 17. Confalonieri M, Aiolfi S, Patrini G, Scartabellati A, Ghio L, Mauri F, et al. [Severe bronchial spasm crises induced by topical administration of eyedrops with timolol base, a non-selective beta blocking agent]. Recenti Prog Med 1991; 82:402-4.
- 18. Odeh M, Oliven A, Bassan H. Timolol eyedrop-induced fatal bronchospasm in an asthmatic patient. J Fam Pract 1991; 32:97-8.
- 19. Le Jeunne CL, Hugues FC, Dufier JL, Munera Y, Bringer L. Bronchial and cardiovascular effects of ocular topical B-antagonists in asthmatic subjects: comparison of timolol, carteolol, and metipranolol. J Clin Pharmacol 1989; 29:97-101.
- 20. Lang DM. Anaphylactoid and anaphylactic reactions. Hazards of beta-blockers. Drug Saf 1995; 12:299-304.
- 21. Cleaveland CR, Rangno RE, Shand DG. A standardized isoproterenol sensitivity test. The effects of sinus arrhythmia, atropine, and propranolol. Arch Intern Med 1972; 130:47-52.

22. Hepner MJ, Ownby DR, Anderson JA, Rowe MS, Sears-Ewald D, Brown EB. Risk of systemic reactions in patients taking beta-blocker drugs receiving allergen immunotherapy injections. J Allergy Clin Immunol 1990; 86:407-11.

- 23. Muller UR, Haeberli G. Use of beta-blockers during immunotherapy for Hymenoptera venom allergy. J Allergy Clin Immunol 2005; 115:606-10.
- 24. Rueff F, Przybilla B, Bilo MB, Muller U, Scheipl F, Aberer W, et al. Predictors of side effects during the buildup phase of venom immunotherapy for Hymenoptera venom allergy: the importance of baseline serum tryptase. J Allergy Clin Immunol 2010; 126:105-11 e5.
- 25. Rueff F, Przybilla B, Bilo MB, Muller U, Scheipl F, Aberer W, et al. Predictors of severe systemic anaphylactic reactions in patients with Hymenoptera venom allergy: importance of baseline serum tryptase-a study of the European Academy of Allergology and Clinical Immunology Interest Group on Insect Venom Hypersensitivity. J Allergy Clin Immunol 2009; 124:1047-54.
- 26. Brown SG. Clinical features and severity grading of anaphylaxis. J Allergy Clin Immunol 2004; 114:371-6.
- 27. Stoevesandt J, Hain J, Kerstan A, Trautmann A. Over- and underestimated parameters in severe Hymenoptera venom-induced anaphylaxis: cardiovascular medication and absence of urticaria/angioedema. J Allergy Clin Immunol 2012; 130:698-704 e1.
- 28. Lee S, Hess EP, Nestler DM, Bellamkonda Athmaram VR, Bellolio MF, Decker WW, et al. Antihypertensive medication use is associated with increased organ system involvement and hospitalization in emergency department patients with anaphylaxis. J Allergy Clin Immunol 2013; 131:1103-8.
- 29. Tunon-de-Lara JM, Villanueva P, Marcos M, Taytard A. ACE inhibitors and anaphylactoid reactions during venom immunotherapy. Lancet 1992; 340:908.
- 30. Ober Al, MacLean JA, Hannaway PJ. Life-threatening anaphylaxis to venom immunotherapy in a patient taking an angiotensin-converting enzyme inhibitor. J Allergy Clin Immunol 2003; 112:1008-9.
- 31. Hermann K, Ring J. The renin angiotensin system and hymenoptera venom anaphylaxis. Clin Exp Allergy 1993; 23:762-9.
- 32. Hermann K, von Tschirschnitz M, Ebner von Eschenbach C, Ring J. Histamine, tryptase, norepinephrine, angiotensinogen, angiotensin-converting enzyme, angiotensin I and II in plasma of patients with hymenoptera venom anaphylaxis. Int Arch Allergy Immunol 1994; 104:379-84.
- 33. Hermann K, Ring J. The renin-angiotensin system in patients with repeated anaphylactic reactions during hymenoptera venom hyposensitization and sting challenge. Int Arch Allergy Immunol 1997; 112:251-6.
- 34. Stoevesandt J, Hain J, Stolze I, Kerstan A, Trautmann A. Angiotensin-converting enzyme inhibitors do not impair the safety of Hymenoptera venom immunotherapy build-up phase. Clin Exp Allergy 2014; 44:747-55.
- 35. Bilo BM, Rueff F, Mosbech H, Bonifazi F, Oude-Elberink JN, Hypersensitivity ElGolV. Diagnosis of Hymenoptera venom allergy. Allergy 2005; 60:1339-49.
- 36. Bonifazi F, Jutel M, Bilo BM, Birnbaum J, Muller U, Hypersensitivity ElGoIV. Prevention and treatment of hymenoptera venom allergy: guidelines for clinical practice. Allergy 2005; 60:1459-70.
- 37. Ring J, Messmer K. Incidence and severity of anaphylactoid reactions to colloid volume substitutes. Lancet 1977; 1:466-9.
- 38. Mueller HL. Diagnosis and treatment of insect sensitivity. J Asthma Res 1966; 3:331-3.